CLINICAL TRIAL: NCT07359261
Title: Transpulmonary Assessment for Individualized Lung Optimization in Patients Living With Obesity Research - Positive End-Expiratory Pressure
Brief Title: Transpulmonary Assessment for Individualized Lung Optimization in Obese Patients
Acronym: TAILOR-PEEP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00154874
Record Dates: First submitted 2026-01-05; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Failure
Keywords: PEEP; obesity; mechanical ventilation
MeSH Terms: conditions — Respiratory Insufficiency; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esophageal-balloon guided (Experimental): Esophageal balloon catheter placed within 4 hours of randomization. PEEP titrated to achieve end-expiratory transpulmonary pressure of 0-2 cmH2O (up to 8 cmH2O for P/F ratio <200). PEEP adjusted in 2 cmH2O increments with 5-minute stabilization periods. Safety limits: transpulmonary driving pressure <15 cmH2O, end-inspiratory transpulmonary pressure <20 cmH2O. Reassessment twice daily (approximately 0800 and 2200). Catheter removed prior to extubation or at 28 days, whichever occurs first.
  Interventions: Procedure: Esophageal pressure-guided PEEP titration
- Standard of Care (Active Comparator): PEEP management according to current standard practice. For patients meeting ARDS criteria, PEEP titrated using the ARDSNet PEEP/FiO2 table. For non-ARDS patients, PEEP titrated per local practice to optimize oxygenation while monitoring hemodynamic tolerance and respiratory mechanics. No esophageal pressure monitoring.
  Interventions: Other: Standard care PEEP management

INTERVENTIONS:
Procedure: Esophageal pressure-guided PEEP titration — PEEP titration guided by transpulmonary pressure measurements using esophageal manometry. Esophageal balloon catheter inserted within 4 hours of randomization, positioned at 35-40 cm depth with position verified by cardiac oscillations and occlusion test. PEEP titrated in 2 cmH2O increments targeting end-expiratory transpulmonary pressure 0-2 cmH2O, with option to target up to 8 cmH2O for severe hypoxemia (P/F <200). Safety limits enforced: transpulmonary driving pressure <15 cmH2O, end-inspiratory transpulmonary pressure <20 cmH2O. Measurements performed twice daily. Catheter removed at extubation or day 28.
  Other Names: Transpulmonary pressure-guided PEEP titration; Pes-guided PEEP management
  Arms: Esophageal-balloon guided
Other: Standard care PEEP management — PEEP management per institutional standard practice without esophageal pressure monitoring. For patients meeting ARDS criteria, PEEP titrated using ARDSNet low PEEP/FiO2 table. For non-ARDS patients, PEEP titrated to optimize oxygenation while monitoring hemodynamic tolerance and respiratory mechanics per treating clinician judgment.
  Arms: Standard of Care

SUMMARY:
This protocol describes a randomized controlled feasibility vanguard study designed to investigate the implementation and effects of esophageal pressure-guided positive end-expiratory pressure (PEEP) titration in patients with high body mass index (BMI) mechanically ventilated patients at the Edmonton Zone. The study will enroll 30 patients with body mass index (BMI) >=30 kg/m2 who require invasive mechanical ventilation, randomizing them in a 1:1 ratio to receive either esophageal pressure-guided PEEP titration or standard care management. The primary objective focuses on establishing the feasibility of conducting a larger definitive trial, while secondary objectives examine differences in applied PEEP levels, respiratory mechanics, and clinical outcomes between groups. The intervention protocol targets end-expiratory transpulmonary pressure of 0-2 cmH2O.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Body mass index ≥30 kg/m²
* Intubated and receiving passive mechanical ventilation
* Within 24 hours of intubation
* Anticipated need for mechanical ventilation for at least 48 hours

Exclusion Criteria:

* Known or suspected esophageal varices
* Esophageal surgery within 3 months
* Known esophageal stricture or perforation
* Active upper gastrointestinal bleeding
* Severe coagulopathy (INR >3.0 or platelet count <30,000/μL)
* Known or suspected intracranial hypertension without intracranial pressure monitoring device demonstrating controlled intracranial pressure (<20 mmHg)
* Severe hemodynamic instability at treating physician discretion
* Known pregnancy
* Moribund state with expected survival <48 hours
* Receiving extracorporeal membrane oxygenation (ECMO)
* Open abdomen post-operatively
* Previous enrollment in this study
* Any other contraindication to esophageal balloon placement as determined by clinical team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of conducting a definitive trial (composite) | 14 months
  Composite feasibility assessment including: (1) Recruitment rate (patients enrolled per month, target 1-1.5/month); (2) Successful esophageal catheter placement rate in intervention arm; (3) Protocol adherence (percentage of scheduled transpulmonary pressure measurements completed, compliance with PEEP titration algorithm); (4) Data completeness for average PEEP over 7 days.

SECONDARY OUTCOMES:
Average PEEP | 7 days
  Key secondary endpoint. Mean positive end-expiratory pressure during mechanical ventilation
Driving Pressure | 7 days
  Difference in driving pressure between groups
Partial oxygen pressure over inspired oxygen fraction ratio | 7 days
  P/F ratio
Days alive and free of mechanical ventilation | Up to hospital discharge assessed up to 30 days
  Days alive and free of mechanical ventilation
Days alive and outside the intensive care unit | Up to hospital discharge assessed up to 30 days
  Days alive and outside the intensive care unit
Hospital Mortality | Up to hospital discharge assessed up to 30 days
  Hospital Mortality
Hemodynamics Instability | Up to 7 days
  Hemodynamics Instability during PEEP Titration defined as a new start of vasopressors at any dose or an increase in vasopressor dose by 20%

OTHER OUTCOMES:
Catheter-related complications | 7 days
  Occurrence of esophageal catheter complications (perforation, bleeding)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - Sturgeon Community Hospital, St. Albert, Alberta

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After publication
Access Criteria: Anonymized data may be shared after discussion with study steering committee, approval from ethics from University of Alberta, and establishment of data sharing agreement.